CLINICAL TRIAL: NCT05725200
Title: Study to Investigate Outcome of Individualized Treatment Based on Pharmacogenomic Profiling & Ex Vivo Drug Sensitivity Testing of Patient-derived Organoids in Patients With Metastatic Colorectal Cancer
Brief Title: Study to Investigate Outcome of Individualized Treatment in Patients With Metastatic Colorectal Cancer
Acronym: EVIDENT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tormod Kyrre Guren, MD, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVIDENT
Record Dates: First submitted 2023-01-06; First posted 2023-02-13 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — alectinib; Cetuximab; Crizotinib; Dasatinib; Everolimus; encorafenib; Gemcitabine; idelalisib; larotrectinib; Methotrexate; palbociclib; Panobinostat; pembrolizumab; Trastuzumab; talazoparib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized treatment in patients with metastatic colorectal cancer (Experimental): Interventions with anti-cancer drugs having marketing authorisation in Norway will be used in this study.
  The intervention will be study drugs as monotherapy or treatment with approved combinations.
  This trial will facilitate access to potentially effective interventions to which they would otherwise not have access.
  Interventions: Drug: Alectinib; Drug: Cetuximab; Drug: Crizotinib; Drug: Dasatinib; Drug: Everolimus; Drug: Encorafenib; Drug: Gemcitabine; Drug: Idelalisib; Drug: Larotrectinib; Drug: Methotrexate; Drug: Palbociclib; Drug: Panobinostat; Drug: Pembrolizumab; Drug: Petrozumab; Drug: Trastuzumab; Drug: Talazoparib; Drug: Venetoclax

INTERVENTIONS:
Drug: Alectinib — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current Summary of Product Characteristics (SMPC) and package Insert.
Drug: Cetuximab — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Crizotinib — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Dasatinib — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Everolimus — Dosage form, dosage, frequency and duration are described in the current SMPC and package Insert.
Drug: Encorafenib — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Gemcitabine — Dosage form, dosage, frequency and duration are described in the current SMPC and package Insert.
Drug: Idelalisib — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Larotrectinib — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Methotrexate — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Palbociclib — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Panobinostat — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Pembrolizumab — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Petrozumab — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Trastuzumab — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Talazoparib — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.
Drug: Venetoclax — Dosage form, dosage, frequency and duration are to be implemented by study investigators as described in the current SMPC and package Insert.

SUMMARY:
The purpose of the study is to investigate the effect and side effects of personalized cancer treatment in patients with metastatic colorectal cancer (bowel cancer). All patients included must have metastatic bowel cancer and receive or have received at least two lines of standard chemotherapy. The cancer must not be available for surgery with curative intent.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate individualized systemic anti-cancer treatment of metastatic colorectal cancer (mCRC), selected by a combined pharmacogenomic drug sensitivity profile with a molecular profiling of the tumor tissue and an ex vivo drug sensitivity testing of patient-derived organoids (PDOs). The combined pharmacogenomic drug sensitivity profile will be provided by Department of Molecular Oncology, Institute for Cancer Research, Oslo University Hospital (OUS) and will be a result of either i) a pre-screening performed in this study or ii) from previous biomarker analyses and drug sensitivity testing of PDOs as part of an ongoing translational research project at Dept. of Molecular Oncology. The combined pharmacogenomic profile will be interpreted by an institutional multidisciplinary tumor board (MTB), and in cases where the MTB strongly suggests that the patient will benefit from one of the interventions offered by this study, the patient will be invited to participate. No formal hypotheses testing will be performed in the study, but it aims to show that it is feasible, in an unselected population of patients with mCRC, to select patients for individualized therapy based on a broad genomic and transcriptomic profiling and ex vivo drug sensitivity testing of cultured PDOs from the patient's own tumor cells, and to provide evidence that a combined pharmacogenomic profile can predict objective antitumor responses to systemic anticancer therapies, including drugs not approved for treatment of patients with mCRC, in the setting of third-line therapy or in later lines. In addition, this study will be part of several translational research projects at the Department of Molecular Oncology.

ELIGIBILITY:
Pre-screening:

Inclusion Criteria:

* Has a histologically-proven locally advanced or metastatic adenocarcinoma from colon or rectum
* Has received or is receiving systemic treatment for mCRC
* Has non-resectable metastases and eligible to undergo a radiological-guided core biopsy from at least one metastasis
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Has measurable or evaluable disease (per RECIST v1.1)
* Is capable of giving signed informed consent, as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

* Has other clinically significant medical conditions which, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or which could jeopardize compliance with study requirements.

MAIN STUDY:

Inclusion Criteria:

1. Has a histologically-proven locally advanced or metastatic adenocarcinoma from colon or rectum (mCRC)
2. Has received at least two lines of SOC chemotherapy for mCRC Note: 1) For patients who develop a metastatic relapse < 6 months after completed total neo-adjuvant treatment in conjunction with a metastasectomy, this treatment will be considered as one line (e.g. first-line) chemotherapy. 2) Patients with the gene RAS wild-type tumors should have received or have been offered and refused prior treatment with antibodies against epidermal growth factor receptor (EGFR) (e.g. in combination with prior lines of chemotherapy) unless it was contraindicated due to underlying conditions or the tumor contains molecular alterations suggested to provide primary resistance to EGFR-targeted therapy.
3. Has full combined pharmacogenomic profile (genomic and transcriptomic profile of the patients tumor and ex vivo drug sensitivity testing of PDOs from the patient's own tumors cells) from which the MTB suggests a treatment with one of the defined targeted anti-cancer therapies provided this study
4. Has measurable or evaluable disease (per RECIST v1.1)
5. ECOG performance status 0 or 1
6. For orally administered drugs, the participant must be able to swallow and tolerate oral medication and must have no known malabsorption syndrome.
7. Because of the risks of drug treatment to a developing fetus, women of child-bearing potential and men must agree to use adequate contraception in accordance with the respective SmPC and as listed in Appendix 4 for the duration of study participation, and up to 7 months following completion of study therapy. Male study patients, even if surgically sterilized, (i.e. post-vasectomy) must agree to one of the following: practice effective barrier contraception during the entire study treatment period and through 6 months after the last dose of study drug, or completely abstain from sexual intercourse.
8. Has acceptable organ function as defined below. However, as noted below (exclusion criterion 16), drug-specific inclusion/exclusion criteria specified in the Appendix 16/respective SmPC for each agent will take precedence for this and all inclusion criteria:

   1. Absolute neutrophil count ≥ 1.5/nL (nL = nano Litre)
   2. Hemoglobin > 10 g/dL
   3. Platelets > 100/nL
   4. Total bilirubin < 1.5 x institutional upper limit of normal (ULN)
   5. Aspartate aminotransferase AST (SGOT) and alanine aminotransferase ALT(SGPT) < 2.5 x institutional upper limit of normal (ULN) (or < 5 x ULN in patients with known hepatic metastases)
   6. Calculated or measured creatinine clearance ≥ 50 mL/min/1.73 m2

Exclusion Criteria:

1. Has ongoing toxicity > CTCAE grade 2, other than peripheral neuropathy and alopecia, related to anti-tumor treatment that was completed within 4 weeks prior to registration. Patients with ongoing peripheral neuropathy of ≥ CTCAE grade 3 will be excluded.
2. Has received previous treatment with the selected study drug for the same malignancy.
3. Has a tumor with a genomic variant known to confer resistance to an anti-cancer agent available in this study, the patient will not be eligible to receive that agent but will be eligible to receive other drugs available in this study if all inclusion and exclusion criteria are met for that drug.
4. Is receiving any other anti-cancer therapies (cytotoxic, biologic, radiation, or hormonal other than for replacement). Participants may be on warfarin, low molecular weight heparin or direct factor Xa inhibitors, unless such therapies are prohibited by drug-specific exclusion criteria (please consult the corresponding SmPC and Appendix 16 for prohibited medication and contraindication/precautions).
5. Is pregnant or breastfeeding or refusing any type of required contraception methods.
6. Has known Central Nervous System (CNS) metastases.
7. Has preexisting cardiac conditions, including uncontrolled or symptomatic angina, uncontrolled atrial or ventricular arrhythmias, or symptomatic congestive heart failure.
8. Has left ventricular ejection fraction (LVEF) known to be < 40%.
9. Has had a stroke (including TIA) or an acute myocardial infarction within 6 months before the first dose of study treatment.
10. Has had acute gastrointestinal bleeding within 1 month of start of treatment
11. Has other clinically significant medical conditions which, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or which could jeopardize compliance with study requirements.
12. Meets any of the assigned drug contraindications or other drug-specific exclusion criteria as described in the respective SmPC and in Appendix 16

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2038-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-Screening: Obtain a combined pharmacogenomic profile which can be used to provide a MTB-nominated treatment | In average of 3 months
  Number of participants that obtain a full combined pharmacogenomic profile which can be used to provide an MTB-nominated treatment in the Main Study.
Main Study: To evaluate the anti-tumor activity, measured as objective response rate (ORR) of MTB-nominated therapies with drugs not approved or implemented in standard of care (SOC) for treatment of mCRC. | Through study completion, in average 6 months
  Number of patients who achieve objective response according RECIST 1.1 in the total study population and each study drug cohort of MTB-nominated therapies with drugs not approved or implemented SOC for treatment of mCRC.

SECONDARY OUTCOMES:
Pre-Screening: To obtain a full combined pharmacogenomic profile from a tumor biopsy that is eligible for treatment decisions in a standard oncology practice. | Through study completion, approximately 4 years
  Pre-Screening:
  Number of participants who achieve a full combined pharmacogenomic profile eligible for treatment decisions either by
  * An MTB-nominated treatment provided in the Main Study
  * An MTB-nominated treatment considered as SOC
  * An MTB-nominated treatment not considered as SOC and not provided in the Main Study
  * No MTB-nominated treatment suggested
Main Study: Progression-free survival (PFS) and duration of response (DOR) | Through study completion, approximately 6 months
  Progression-free survival (PFS) and duration of response (DOR) by RECIST 1.1, of participants receiving an MTB-nominated anti-cancer therapy, by calculation of number of days, weeks or years.
Main Study: Overall survival (OS) | Through study completion, approximately 6 months
  OS of participants receiving MTB-nominated anti-cancer therapy, defined as the time from first dose of MTB-nominated treatment to date of death from any cause by calculation of number of days, weeks or years.
Main Study: Safety and tolerability of the different MTB-nominated treatments | Through study completion, approximately 6 months
  Register adverse events (AE) in accordance with CTCAE v 5.1
Main Study: Objective response of an MTB-nominated anti-cancer therapy compared to objective response to the prior line(s) SOC treatment. | Through study completion, approximately 6 months
  Number of patients who achieve objective response according to RECIST 1.1 from anti-cancer therapy (SOC) in prior lines.
Main Study: Efficacy of MTB-nominated anti-cancer therapy compared to the efficacy of prior lines SOC treatment. | Through study completion, approximately 6 months.
  DOR and PFS by RECIST 1.1 of participants receiving an MTB-nominated treatment and from anti-cancer therapy received in prior lines of SOC in each patient, by calculation of number of days, weeks or years.
Main study: Objective response of an MTB-nominated anti-cancer therapy compared to objective response to the next line(s) SOC treatment. | Through study completion, approximately 6 months.
  Number of patients who achieve objective response according to RECIST 1.1 from receiving anti-cancer therapy in the next/later lines.
Main study: Efficacy of an MTB-nominated anti-cancer therapy compared to the efficacy achieved by the next line(s) of SOC treatment. | Through study completion, approximately 6 months.
  DOR and PFS by RECIST 1.1 of participants receiving an MTB-nominated treatment and from anti-cancer therapy in the next/later lines of SOC treatment in each patient, by calculation of number of days, weeks or years.
Main study: Patient-reported outcome measures. | Through study completion, approximately 6 months.
  Describe patient-reported quality of life during the MTB-nominated treatment, registered by EORTC Quality of Life Questionnaire (QLQ)-C30 questionnaire.
  The EORTC QLQ-C30 questionnaire consisted of 30 questions generating five functional scores (physical, role, cognitive, emotional, and social); a global health status/global quality of life scale score; three symptom scale scores (fatigue, pain, and nausea and vomiting); and six stand alone one-item scores that capture additional symptoms (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) and perceived financial burden. All the scales and single-item scores were linearly transformed so that each score ranged from 0 to 100. A higher score on the global health and functioning subscales is indicative of better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Tormod K Guren, MDPhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway